CLINICAL TRIAL: NCT03586193
Title: Application of Pars Plana Vitrectomy in the Treatment of Macular Schisis in High Myopic Eyes
Brief Title: Pars Plana Vitrectomy Alone in the Treatment of Macular Schisis in High Myopic Eyes
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aier School of Ophthalmology, Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: SHIRB2018014
Record Dates: First submitted 2018-06-15; First posted 2018-07-13 (Actual); Last update posted 2018-07-13 (Actual); Status verified 2018-07

CONDITIONS: Retinal Disease; Macular Retinoschisis
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients with HMF: Patients who are diagnosed as high myopic macular schisis and agree to receive pars plana vitrectomy as the treatment are planned to allocated in this group
  Interventions: Procedure: Pars plana vitrectomy

INTERVENTIONS:
Procedure: Pars plana vitrectomy — pars plana vitrectomy without ICG staining and ILM peeling

SUMMARY:
High myopic schisis (HMF) has the clinical feature of separation between retinal layers. It is sometimes accompanied with foveal retinal detachment, macular lamellar hole, epiretinal membrane and vitreous retraction. HMF may develop to macular hole, macular detachment and will damage the visual function. Pars plana vitrectomy (PPV) is a commonly used surgery in the treatment of HMF. PPV together with internal limiting membrane (ILM) peeling and long-term gas tamponade was reported to be safe and effective. But nowadays there was no available long-term gas in our country. Also, whether ILM peeling is necessary remains controversial, Indole cyanine green (ICG)was proved to have potential toxicity to the retina and the ILM peeling has the risk of causing secondary macular hole. We propose to make a prospective nonrandomized controlled study to evaluate the safety and efficiency of using PPV alone in the treatment of HMF.

ELIGIBILITY:
Inclusion Criteria:

1. Patients diagnosed as high myopic macular retinoschisis, with axial length more than 26.5mm.
2. Morphologic manifestation in OCT shows split between retinal layers in macular area.
3. Patients without severe systemic disease and can tolerate surgery.

Exclusion Criteria:

1. Patients also have other ocular disease, including glaucoma, keratitis,uveitis, retinal detachment,etc.
2. Patients with nystagmus or have difficult to open the eye.
3. Patients with severe systemic disease and cannot tolerate surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Study population will be selected from the in-patients in Shanghai Aier Eye Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-05-31 (Estimated)

PRIMARY OUTCOMES:
The morphologic change of macular area | OCT will be done one day before surgery and one week, one month, three months and six months after surgery
  The thickness of the macular fovea in optical coherence tomography (OCT)

SECONDARY OUTCOMES:
The best corrected visual acuity (BCVA) change | One day before surgery and one week, one month, three months and six months after surgery
  The BCVA of all involved patients
The best corrected near visual acuity (BCNVA) change | One day before surgery and one week, one month, three months and six months after surgery
  The BCNVA of all involved patients
The visual function change | One day before surgery and one week, one month, three months and six months after surgery
  The contrast sensitivity of all involved patients

CONTACTS AND LOCATIONS:
Overall Officials: Wensheng Li, Doctor, Study Director — Shanghai Aier Eye Hospital
Locations (1):
- Shanghai Aier Eye hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: After this study is finished the data will become available for 1year.
Access Criteria: The analytical data will be accessed in published articles.

REFERENCES:
- [Background] Chang JS, Flynn HW Jr, Engelbert M, Shane AR, Smiddy WE, Chang S. Pars plana vitrectomy in patients with myopic macular retinoschisis. Br J Ophthalmol. 2014 Apr;98(4):534-7. doi: 10.1136/bjophthalmol-2013-304578. Epub 2014 Jan 10. PMID 24414402
- [Result] Zhang Z, Wei Y, Jiang X, Zhang S. PARS PLANA VITRECTOMY AND WIDE INTERNAL LIMITING MEMBRANE PEELING WITH PERFLUOROPROPANE TAMPONADE FOR HIGHLY MYOPIC FOVEOSCHISIS-ASSOCIATED MACULAR HOLE. Retina. 2017 Feb;37(2):274-282. doi: 10.1097/IAE.0000000000001146. PMID 27429390
- [Result] Rey A, Jurgens I, Maseras X, Carbajal M. Natural course and surgical management of high myopic foveoschisis. Ophthalmologica. 2014;231(1):45-50. doi: 10.1159/000355324. Epub 2013 Nov 12. PMID 24246446